CLINICAL TRIAL: NCT02522182
Title: ALLiance for sEcondary PREvention After an Episode of Acute Coronary Syndrome. The ALLEPRE Trial: a Fully Nurse-led Intensive Intervention Programme
Brief Title: ALLiance for sEcondary PREvention After an Episode of Acute Coronary Syndrome (ALLEPRE)
Acronym: ALLEPRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Diego Ardissino, MD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E35E09000880002
Record Dates: First submitted 2015-07-21; First posted 2015-08-13 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2023-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiovascular Secondary Prevention; Nurse's Role
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Secondary Prevention Programme (Experimental): The Nurse-led Intensive Secondary Prevention Programme consists of programmed 9 sessions involving the trained nurses and the patients randomised to the experimental programme: before discharge, and one, three, six, 12, 18, 24, 36 and 48 months follow up. During the sessions the nurse will record the main clinical parameters (risk factors, lifestyle habits, adherence to therapy, psychological characteristics), any discrepancies between patient reports and the recommended goals and then activate the interventions in order to correct the discrepancies. The activation of the pre-established multidisciplinary network (anti-smoking, anti-diabetes and anti-hypertension centres, and psychological support) is completely under the nurses' control.
  Interventions: Behavioral: Nurse-led Intensive Secondary Prevention Programme
- Usual Treatment (Active Comparator): The patients randomised to the control group will follow the Usual Treatment for secondary prevention of the hospital to which they were admitted
  Interventions: Behavioral: Usual Treatment

INTERVENTIONS:
Behavioral: Nurse-led Intensive Secondary Prevention Programme — Information related to intervention description have been already included in arm/group description
  Arms: Intensive Secondary Prevention Programme
Behavioral: Usual Treatment — Information related to intervention description have been already included in arm/group description
  Arms: Usual Treatment

SUMMARY:
The purpose of the ALLEPRE trial is to compare the benefit offered by a structured, intensive and fully nurse-led intensive secondary prevention intervention programme with that offered by standard of care in a high-risk population of patients admitted to hospital because of an ACS.

DETAILED DESCRIPTION:
ALLEPRE enrols a population of residents in Emilia Romagna with a diagnosis of ACS (unstable angina, non-ST segment elevation myocardial infarction, ST segment elevation myocardial infarction) who were admitted to the specialist cardiological departments of the participating centres up to 20 days after the index event.

All eligible patients are randomised 1:1 to the nurse-led intensive secondary prevention programme (ISPP: intervention/experimental arm) or usual treatment (UT: control arm).

Randomisation is centralised by means of IVRS under the responsibility of the Study Coordinator and the Principal Investigator at each hospital centre, and the patients are the allocated to groups by e-mail. Due to the nature of the study, neither participants nor research personnel can be blinded to the group assignments. The randomisation data are kept at the coordinating centre.

OPERATIVE PHASE After randomisation, all of the patients in both arms undergo a baseline examination and are required to return to their reference centre for follow-up visits after 12, 24 and 60 months for outcome assesment. Outcomes will also be recorded after 36 and 48 months on the basis of telephone enquiries.

ISPP: intervention arm. This consists of a series of programmed sessions involving the centrally trained nurses and the patients randomised to the ISPP. There will be a total of nine sessions: before discharge, and one, three, six, 12, 18, 24, 36 and 48 months after discharge. During the sessions, each of which will last for about one hour, the trained nurse will record the main clinical parameters (i.e. risk factors, lifestyle habits, adherence to therapy, and any discrepancies between patient reports and the recommended goals) using an ad hoc clinical file (SIM: scheda infermieristica multidimensionale or multidimensional nursing form), and then activate the interventions laid down by the pre-specified rules inside the SIM in order to correct the discrepancies. The activation of the pre-established multidisciplinary network (anti-smoking, anti-diabetes and anti-hypertension centres, and psychological support) is completely under the nurses' control.

Caregivers are encouraged to support the patients in achieving behavioural changes over time.

Adherence to the proven secondary prevention treatments is monitored using the Morisky scale in order to ensure that each of the following classes of cardioprotective medications are prescribed according to the guidelines at the doses used in clinical trials: antiplatelet therapy, beta-blockers, angiotensin-converting enzyme inhibitors or angiotensin II receptor blockers, and statins. The reasons for non-adherence also investigated in order to ensure more targeted interventions. The risk factor and lifestyle behaviour goals are to stop smoking, eat a healthy Mediterranean diet, undertake physical activity for at least 30 minutes/day on five days/week, and maintain a body mass index (BMI) of <25 kg/m2, systolic blood pressure of <140, LDL cholesterol levels of <70 mg/dL (1.81 mmol/L). A further goal for all diabetic subjects is good glycemic control.

The nurses also assess the subjects' psychological characteristics by means of a questionnaire that measures anxiety, depression, anger and hostility, type A and type D personality, perceived social support and perceived self-efficacy, and use an ad hoc questionnaire for referral to a psychologist if necessary.

To ensure the same nurse intervention in all partecipating centers the study started with a preliminary TRAINING PHASE involving professional nurses proposed by the participating centres (6-10 per centre, 50% from a hospital setting, 50% from a community setting). The training programme was coordinated by the Training and Continuous Education Centre of Parma University Hospital, and delivered by a multidisciplinary team of medical/nursing/psychological experts with the aid of ad hoc paper-based teaching materials. It consisted of three 8-hour sessions held on consecutive days during which the nurses were trained in secondary CVD prevention and how to take multi-dimensional and structured responsibility for ACS patients using appropriate communication strategies aimed at reducing risk factors, modifying lifestyles and improving adherence to prescribed pharmacological therapy. The programme was repeated four times in order to allow the creation of small groups (20 participants) and better interactions.

UT: control arm. The patients randomised to the control group will follow the standard for secondary prevention of the hospital to which they were admitted.

DATA MANAGEMENT All of the data are peripherally recorded in electronic case report forms and stored for further analysis. An external monitoring provides for all partecipating centrers the clinical data verification, the accuracy and the completeness of electronic case report forms.

Sample size and statistical aspects On the basis of the results of the GRACE UK-Belgian Study, it is conservatively expected that the cumulative rate of clinical endpoints in the standard care arm (cardiovascular mortality, non-fatal reinfarction, non-fatal stroke) during the five years' follow-up will be 28%. Using the formula of Lakatos and Lan (Statistics in Medicine, 1992), in order to detect a 25% risk reduction in the experimental group, with 90% power and a two-sided significance level of 0.25, at least 1030 patients are required in each group.

However, a two-year interim analysis of the major clinical endpoint will show the real divergence of the curves and provide further information for estimating the required duration of the study more precisely. The estimated sample size is also valid for the analysis of the first primary endpoint.

The plan of the primary and secondary analyses includes a Kaplan-Meier analysis of the time to an event, the HR, and log-rank comparisons based on the ITT and PP populations.

The baseline characteristics of the intervention and control group will be compared using the chi-squared test for categorical factors and Student's t test for independent samples for continuous factors. The data will be expressed as mean values ± standard deviations. All of the statistical analyses will be made using the SPSS programme.

A secondary heterogeneity analysis of the primary clinical outcomes will be made by stratifying the patients by age, sex, center, literacy level, diabetes, hypertension, smoking habits, family history, type of myocardial infarction (STEMI vs NSTEMI), and hospital characteristics. Analysis of repeated measures will be used to evaluate the changes in the primary surrogate end point over time.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients aged >18 years with an ACS (unstable angina, non- ST-segment elevation myocardial infarction [MI], or ST-segment elevation MI [International Classification of Diseases, Ninth Revision, Clinical Modification codes 41071, 41001, 41011, 41021, 41031, 41041, 41051,41061, 41081, and 41091]) who are admitted to the Cardiological Divisions of the 6 participating centers in Emilia-Romagna (Italy) are considered for enrolment for up to 20 days after the index event and before being discharged.

Exclusion Criteria:

Once it has been verified that the patients are capable of participating in a prospective study, the only exclusion criterion is a life expectancy of b12 months because of a severe noncardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2060 (Actual)
Dates: Start 2012-10; Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to the goals of classic cardiovascular risk factors:
  - number of patients (nop) with systolic blood pressure <140 mmHg, divided by total nop.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to the goals of classic cardiovascular risk factors:
  - nop with LDL cholesterol <70 mg/dL, divided by total nop.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to the goals of classic cardiovascular risk factors:
  - number of non-smokers, divided by the total nop.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to the goals of classic cardiovascular risk factors:
  - nop with HbAC1 <7%, divided by total nop.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  The number of patients with the target body mass index (18-24.9) divided by the total nop.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to life style modifications:
  - Number of patients eating at least 5 servings friut/vegetable/day divided by total nop at month 24.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  The number of patients eating at least 2 fish servings/wk divided by the total
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to life style modifications:
  The number of patients spending at least 30 min/d, 5 times/wk on recreational exercise divided by the total number of patients.
The difference in the degree of adherence to the goals concerning risk factors, lifestyle modifications and pharmacological therapy. | 24 months
  Adherence to medications:
  The number of patients with a high degree of adherence to medications (Morisky Medication Adherence Scale score 3-4) divided by the total nop.
Major adverse events | 5 years
  Composite of cardiovascular mortality, non-fatal reinfarction, non-fatal stroke

SECONDARY OUTCOMES:
Clinical endpoints | 5 years
  a composite of cardiovascular mortality, nonfatal reinfarction, and nonfatal troke and myocardial ischemia-driven revascularization.
Clinical endpoints | 5 years
  non-fatal reinfarction
Clinical endpoints | 5 years
  non-fatal stroke
Clinical endpoints | 5 years
  cardiovascular mortality
Clinical endpoints | 5 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Diego Ardissino, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (7):
- Italy (7):
  - Ospedale di Baggiovara, Baggiovara, Modena
  - Ospedale Ramazzini di Carpi, Carpi, Modena
  - Ospedale di Vaio, Fidenza, Parma
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza, Piacenza
  - Ospedale Sant'Anna, Castelnovo ne' Monti, Reggio Emilia
  - Ospedale Civile di Guastalla, Guastalla, Reggio Emilia

REFERENCES:
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. Lancet. 2009 Mar 14;373(9667):929-40. doi: 10.1016/S0140-6736(09)60330-5. PMID 19286092
- [Background] Fox KA, Carruthers KF, Dunbar DR, Graham C, Manning JR, De Raedt H, Buysschaert I, Lambrechts D, Van de Werf F. Underestimated and under-recognized: the late consequences of acute coronary syndrome (GRACE UK-Belgian Study). Eur Heart J. 2010 Nov;31(22):2755-64. doi: 10.1093/eurheartj/ehq326. Epub 2010 Aug 30. PMID 20805110
- [Background] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889
- [Background] Wood DA, Kotseva K, Connolly S, Jennings C, Mead A, Jones J, Holden A, De Bacquer D, Collier T, De Backer G, Faergeman O; EUROACTION Study Group. Nurse-coordinated multidisciplinary, family-based cardiovascular disease prevention programme (EUROACTION) for patients with coronary heart disease and asymptomatic individuals at high risk of cardiovascular disease: a paired, cluster-randomised controlled trial. Lancet. 2008 Jun 14;371(9629):1999-2012. doi: 10.1016/S0140-6736(08)60868-5. PMID 18555911
- [Background] Giannuzzi P, Temporelli PL, Marchioli R, Maggioni AP, Balestroni G, Ceci V, Chieffo C, Gattone M, Griffo R, Schweiger C, Tavazzi L, Urbinati S, Valagussa F, Vanuzzo D; GOSPEL Investigators. Global secondary prevention strategies to limit event recurrence after myocardial infarction: results of the GOSPEL study, a multicenter, randomized controlled trial from the Italian Cardiac Rehabilitation Network. Arch Intern Med. 2008 Nov 10;168(20):2194-204. doi: 10.1001/archinte.168.20.2194. PMID 19001195
- [Background] Jorstad HT, von Birgelen C, Alings AM, Liem A, van Dantzig JM, Jaarsma W, Lok DJ, Kragten HJ, de Vries K, de Milliano PA, Withagen AJ, Scholte Op Reimer WJ, Tijssen JG, Peters RJ. Effect of a nurse-coordinated prevention programme on cardiovascular risk after an acute coronary syndrome: main results of the RESPONSE randomised trial. Heart. 2013 Oct;99(19):1421-30. doi: 10.1136/heartjnl-2013-303989. Epub 2013 Jun 28. PMID 23813851
- [Background] de Lorgeril M, Salen P, Martin JL, Monjaud I, Delaye J, Mamelle N. Mediterranean diet, traditional risk factors, and the rate of cardiovascular complications after myocardial infarction: final report of the Lyon Diet Heart Study. Circulation. 1999 Feb 16;99(6):779-85. doi: 10.1161/01.cir.99.6.779. PMID 9989963
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] EUROASPIRE I and II Group; European Action on Secondary Prevention by Intervention to Reduce Events. Clinical reality of coronary prevention guidelines: a comparison of EUROASPIRE I and II in nine countries. EUROASPIRE I and II Group. European Action on Secondary Prevention by Intervention to Reduce Events. Lancet. 2001 Mar 31;357(9261):995-1001. doi: 10.1016/s0140-6736(00)04235-5. PMID 11293642